CLINICAL TRIAL: NCT07298499
Title: Post-Market Clinical Follow-Up of Hearing Aids and Tinnitus Masker Technology
Brief Title: Amplification and Tinnitus Masker Performance and Benefit for Adults With Hearing Loss and Tinnitus
Acronym: StarkeyPMCF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Starkey Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StarkeyPMCF2025; PMCF2025 (Other: Starkey HQ)
Record Dates: First submitted 2025-02-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hearing Aid; Tinnitus
Keywords: hearing aid benefit
MeSH Terms: conditions — Tinnitus | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: The participants will have seven lab sessions and six field trials. In the first session, every participant will be fitted with commercially available, post-market prescription hearing aids. Participants will have follow-up sessions after two, six, twelve, eighteen, and twenty-four weeks. The primary safety outcome measure will be gathered at each session. The primary performance outcome measure will be gathered at the initial session. The primary benefit outcome measures pertaining to the benefit of amplification will be gathered at baseline, at twelve weeks, and at twenty-four weeks, and the primary benefit outcome measures pertaining to tinnitus outcomes will be gathered at each session. At the twelve-week session, participants will be fitted with a tinnitus masker using the same commercially available, post-market prescription hearing aids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Amplification with or without masker (Experimental): Amplification alone or amplification plus tinnitus masker
  Interventions: Device: Hearing Aid; Device: Tinnitus Masker

INTERVENTIONS:
Device: Hearing Aid — Inclusion of hearing aid or not for listening
Device: Tinnitus Masker — Inclusion of tinnitus masker in device

SUMMARY:
This study is a Post-Market Clinical Investigation whose primary purpose is to evaluate hearing aid amplification and tinnitus masker performance for individuals with hearing loss and tinnitus. There are two primary hypotheses that will be assessed in this study:

The use of well-fit amplification alone improves participants' ability to hear and improves tinnitus symptoms as compared to unaided conditions.

The use of well-fit amplification in conjunction with a tinnitus masker improves participants' ability to hear and improves tinnitus symptoms as compared to unaided conditions.

Participants will be fit with hearing aids for 6 months and a tinnitus masker will be activated at the 3-month mark of the study. Outcome measures will evaluate device performance and participant benefit from the devices throughout the study duration.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate hearing aid amplification and tinnitus masker performance, and clinical benefit for adults with hearing loss and tinnitus. The participants of the study will include approximately 100 adults with bilateral hearing loss ranging from mild to profound and mild to severe tinnitus as determined by the Tinnitus Handicap Inventory.

Participants will be fit with hearing aids by a licensed research audiologist. Hearing aid fittings will be verified using real-ear measurements and performance will be evaluated by the response accuracy compared to hearing aid prescriptive targets. Participants will first be fit with only amplification for 3 months. The participants will wear the hearing aids regularly in the field and return to the research facility at several intervals to complete measures of hearing aid performance and listening tasks.

At the three-month mark, a tinnitus masker will be turned on through the participant's hearing aids. The masker will be adjusted to participant preferences for sound quality and masker output will be captured using real-ear measurements. The participants will then wear the hearing aids with a tinnitus masker enabled for 3 months and return to the research facility at several intervals to complete measures of hearing aid performance and listening perception tasks.

Through this study the following hypotheses will be tested:

The use of well-fit amplification alone improves participants' ability to hear and improves tinnitus symptoms as compared to unaided conditions.

The use of well-fit amplification in conjunction with an ear-level tinnitus masker improves participants' ability to hear and improves tinnitus symptoms.

According to the American Speech, Language, and Hearing Association, "fitting and monitoring the use of tinnitus maskers, hearing aids, or other ear-level sound generators" are all acceptable management techniques for tinnitus. However, there is not guidance on the order of management strategies. In the ASHA guidance and peer-reviewed literature, there is no evidence of patient characteristics that indicate the patient will benefit from one intervention over another. There is previous research that indicates well- fit hearing aids providing amplification alone improves tinnitus symptoms in individuals with hearing loss and tinnitus. Widely accepted tinnitus management programs -- Tinnitus Retraining Therapy, Progressive Tinnitus Management, and Tinnitus Activities Treatment-- recommend the use of tinnitus masking devices in addition to amplification as a component of tinnitus management for individuals with hearing loss and tinnitus . In randomized controlled studies, it has been found that participants with tinnitus showed equal improvement with tinnitus symptoms when fit with amplification only and when fit with amplification and sound masker devices when compared to no intervention. These studies indicate improvement in tinnitus with intervention versus no intervention. The present study will continue this line of research with participants wearing hearing aids with amplification alone and hearing aids with amplification and a tinnitus masker.

For this study, all participants will first be fit with hearing aids providing amplification only for 3 months and then the tinnitus masker will be enabled in the hearing aids for the second half of the study. This study design was chosen due to the inability to blind the participant or researcher from the intervention and because it mimics many patients' experiences with clinical protocols. The study design also reduces the potential ethical concern of providing the tinnitus masker and removing it as the researchers may be withholding an effective tinnitus management tool after the participant has already grown accustomed to it. When the tinnitus masker is enabled at the 3-month mark, the participants will continue to have access to an amplification only program they can navigate to with their hearing aids. The participants will be encouraged to remain in the tinnitus masker program as much as possible.

The study hypotheses will be tested by comparing clinical benefit questionnaires against normative data or quantifying minimal clinically important differences from unaided to aided conditions for individual participants. Performance of amplification and tinnitus maskers will be verified using real-ear measurements and will confirm the safety of the hearing aids and tinnitus maskers by following the participants for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old

Native English speaking (defined that all education was done in English)

Bilateral hearing impairment ranging from mild to profound

Mild to severe tinnitus

Ability to commute to research facility

Exclusion Criteria:

* Participants will be advised to consult promptly a doctor, preferably an ear specialist such as an ENT, prior to being fit with the study devices, if they display any of the following conditions:

Visible deformity of the ear, either congenital or traumatic

Fluid, pus, or blood coming out of the ear within the previous 6 months

Pain or discomfort in the ear

History of excessive ear wax or suspicion that something is in the ear canal

Dizziness, either recent or long-standing

Sudden, quickly worsening, or fluctuating hearing loss within the previous 6 months

Hearing loss or ringing (tinnitus) only in one ear or a noticeable difference in hearing between ears

Audiometric air-bone gap equal to or greater than 15 dB at 500 Hz, 1000 Hz, and 2000 Hz

Cognitive impairment

Tinnitus with a somatic origin indicating a need for medical treatment

Current user of noise masker delivered via a wearable device

Hyperacusis or extreme sensitivity to sounds

Is employed by the study sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Provision of adequate amplification | The time frame of this data collection is at the hearing aid fitting which occurs at the initial fitting (Session 1, day 1). This will occur the first time the participant is seen for the study visits.
  Real-ear measures (level of sound at various frequencies measured at the tympanic membrane) will be used to show the hearing aid is providing adequate amplification to compensate for the hearing loss in agreement with a prescriptive fitting formula. The hearing aid responses were measured, and target matched using the Audioscan Verifit system with the ISTS stimuli at various presentation levels (50, 65, and 80 dB SPL). The clinical standard expects measured levels to fall within 5 dB of prescriptive gain targets at 500, 1000, and 2000 Hz, and 8 dB of prescriptive gain targets for 3000 and 4000 Hz.
Device Oriented Subjective Outcome (DOSO) questionnaire to evaluate perceived benefit | The time frame of this data collection will occur at session 3 (6 weeks), session 4 (12 weeks), and session 7 (24 weeks)
  The Device Oriented Subjective Outcome (DOSO) Scale is used to determine the effectiveness of hearing aids in various situations. This questionnaire is answered by the participant in reflection of their experience with hearing aids. Responses to the questionnaire are based upon the participant's perception of their experience with the hearing aids. The DOSO score is numerical and a higher number corresponds to higher satisfaction between 1 and 7.
Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire | The time frame of this data collection will occur at session 1(initial fitting, day 1), session 3 (6 weeks), session 4 (12 weeks), and session 7 (24 weeks)
  The Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire is a widely used measure of hearing aid benefit in a variety of real-life situations. The APHAB is a self-report questionnaire that relies on the participant's perception of their experiences both without hearing aids and after being fit with hearing aids. Scores are numeric between 0 and 100, and difference in score between unaided and aided shows how much of a change is associated with the amplification. Positive numbers mean the amplification provides benefit, while negative numbers mean the amplification is degrading performance.
Tinnitus Handicap Inventory (THI) questionnaire | The time frame of this data collection will occur at session 1 (initial fitting, day 1), session 4 (12 weeks), and session 7 (24 weeks)
  The Tinnitus Handicap Inventory is a widely used questionnaire to understand the impact of tinnitus on someone's daily life. A numeric score is generated between 0 and 100, and the higher the number, the more handicap is generated by the Tinnitus. A change in score between unaided and aided would show either an increase in handicap or decrease in handicap between unaided and aided conditions.
Tinnitus Functional Index (TFI) questionnaire | This data will be collected at Session 1(day 1), Session 2 (2 weeks), Session 3 (6 weeks), Session 4 (12 weeks), Session 5 (14 weeks), Session 6 (18 weeks), Session 7 (24 weeks).
  The Tinnitus Functional Index is a widely used questionnaire to understand the multiple domains of tinnitus severity. The outcome is a numeric value between 0 and 100 corresponding to how well the listener can function in various listening situations. The higher number corresponds to increased difficulty functioning, and comparison between unaided and aided conditions determines how much the aided condition improves functioning.
Monitoring of Treatment-Related Adverse Events as Assessed by Otoscopy | This data will be collected at Session 1(day 1), Session 2 (2 weeks), Session 3 (6 weeks), Session 4 (12 weeks), Session 5 (14 weeks), Session 6 (18 weeks), Session 7 (24 weeks).
  Otoscopy and visual inspection will be conducted at each laboratory visit to examine the structures of the ear that come in contact with the hearing aid, namely the outer ear and the external auditory canal, to look for signs of rubbing, abrasion, or skin reactions which should not occur. Adverse events such as these skin changes or reactions associated with the use of the hearing aids, observed in the study will be reviewed, recorded, and treated according to recommended treatment guidelines to confirm that the devices are not negatively causing soreness or irritation and that the benefits from the devices with respect to hearing and tinnitus outweigh the risks.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hicks, Ph.D., Principal Investigator — VP Education and Audiology
Locations (1):
- Starkey Satellite Research Facility Affordable Hearing Centers 6821 W 120th Ave Ste 2H, Broomfield, CO 80020, Broomfield, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tinnitus Retraining Therapy Trial Research Group; Scherer RW, Formby C. Effect of Tinnitus Retraining Therapy vs Standard of Care on Tinnitus-Related Quality of Life: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2019 Jul 1;145(7):597-608. doi: 10.1001/jamaoto.2019.0821. PMID 31120533
- [Background] Newman CW, Jacobson GP, Spitzer JB. Development of the Tinnitus Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1996 Feb;122(2):143-8. doi: 10.1001/archotol.1996.01890140029007. PMID 8630207
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Jastreboff PJ, Jastreboff MM. Tinnitus Retraining Therapy (TRT) as a method for treatment of tinnitus and hyperacusis patients. J Am Acad Audiol. 2000 Mar;11(3):162-77. PMID 10755812
- [Background] Beck JE, Zaugg TL, Egge JL, Lima EN, Thielman EJ. Progressive Tinnitus Management at Two Veterans Affairs Medical Centers: Clinical Implementation With Modified Protocols. Am J Audiol. 2019 Apr 22;28(1S):162-173. doi: 10.1044/2018_AJA-TTR17-18-0040. PMID 31022363
- [Background] Myers PJ, Griest S, Kaelin C, Legro MW, Schmidt CJ, Zaugg TL, Henry JA. Development of a progressive audiologic tinnitus management program for Veterans with tinnitus. J Rehabil Res Dev. 2014;51(4):609-22. doi: 10.1682/JRRD.2013.08.0189. PMID 25144174
- [Background] Jastreboff PJ. Tinnitus retraining therapy. Prog Brain Res. 2007;166:415-23. doi: 10.1016/S0079-6123(07)66040-3. PMID 17956806
- [Background] Del Bo L, Ambrosetti U. Hearing aids for the treatment of tinnitus. Prog Brain Res. 2007;166:341-5. doi: 10.1016/S0079-6123(07)66032-4. PMID 17956798
- [Background] Cox RM, Alexander GC, Xu J. Development of the Device-Oriented Subjective Outcome (DOSO) scale. J Am Acad Audiol. 2014 Sep;25(8):727-36. doi: 10.3766/jaaa.25.8.3. PMID 25380119
- [Background] Cox RM, Alexander GC. The abbreviated profile of hearing aid benefit. Ear Hear. 1995 Apr;16(2):176-86. doi: 10.1097/00003446-199504000-00005. PMID 7789669
- [Background] Preferred Practice Patterns for the professions of speech-language pathology and audiology. American Speech-Language-Hearing Association. ASHA Suppl. 1993 Mar;35(3 Suppl 11):i-viii, 1-102. No abstract available. PMID 8097652